CLINICAL TRIAL: NCT02106468
Title: The Efficacy of Omega-3 in Treatment of Atrophic/Erosive Lichen Planus and Improvement of Quality of Life: A Randomized, Double Blind, Controlled Study
Brief Title: The Efficacy of Omega-3 in Treatment of Atrophic/Erosive Lichen Planus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Enas Elgendy, Lecuture, October 6 University, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Elgendy - 1
Record Dates: First submitted 2014-03-21; First posted 2014-04-08 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2014-03

CONDITIONS: Oral Lichen Planus
Keywords: Oral Lichen Planus; Corticosteroid; Omega -3
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- prednisone 50 mg tablet (Active Comparator): This group included 15 patients who received prednisone (Delta-cortene Fort®, Lepetit, Carmano, Melano, Italy) at 40mg /day (8 tablets/day in divided dose , 4 tablet at morning and 4 at evening) for 6 weeks then 20mg/day for 2 week then to 10 mg/day for 2 week, and finally to 5 mg /day for the last 2 weeks.
  Interventions: Drug: Prednisone tablet 5mg
- Omega-3 capsules 1000 mg (Active Comparator): This group included 15 patients who received Omega-3 soft gelatin capsules 1000 mg (Super Omega; Technopharma, Cairo, Egypt). The patients received instruction to take one capsule three times daily for 3 months.
  Interventions: Drug: Omega-3 soft capsules 1000 mg

INTERVENTIONS:
Drug: Prednisone tablet 5mg — This group included 15 patients who received prednisone (Delta-cortene Fort®, Lepetit, Carmano, Melano, Italy) at 40mg /day (8 tablets/day in divided dose , 4 tablet at morning and 4 at evening) for 6 weeks then 20mg/day for 2 week then to 10 mg/day for 2 week, and finally to 5 mg /day for the last 2 weeks.
  Other Names: Delta-cortene Fort®, Lepetit, Carmano, Melano, Italy
  Arms: prednisone 50 mg tablet
Drug: Omega-3 soft capsules 1000 mg — This group included 15 patients who received Omega-3 soft gelatin capsules 1000 mg (Super Omega; Technopharma, Cairo, Egypt). The patients received instruction to take one capsule three times daily for 3 months.
  Other Names: Super Omega; Technopharma, Cairo, Egypt
  Arms: Omega-3 capsules 1000 mg

SUMMARY:
This study was initiated to evaluate the potential of dietary supplementation of omega-3 for providing an inexpensive, safe and effective therapeutic agent for managing atrophic/erosive lichen planus.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of OLP (Presence of painful and atrophic-erosive oral Lesions, bilateral, mostly symmetrical lesions, presence of lace-like network of slightly raised white lines).
2. Age between 30-60 years
3. Ability to complete the present clinical trial.

Exclusion Criteria:

1. Pregnant or breast feeding women (pregnancy test for women of child bearing age).
2. Lichenoid reactions caused by certain drugs or dental amalgam.
3. Therapy for oral lichen planus (OLP) in the 6 months prior to the study.
4. Patient doesn't have hepatitis C [after the patients' medical histories were recorded, the patients were given hepatic screening as published elsewhere. 2
5. Presence of candidiasis before treatment.
6. Patients with pre-existing diabetes or an initial random glucose level exceeding 200 mg/dL before initiating steroid therapy were excluded.
7. Hypertensive patients
8. Contraindications for corticosteroid use (immunodeficiency or severe heamatological alterations).

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-05; Primary Completion 2014-06 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Improve quality of the life (Oral Health Impact Profile) | 6 months
  Improve quality of the life was recorded at baseline, 3 and 6 months after treatment.

SECONDARY OUTCOMES:
Size and types (atrophic/erosive) of the lesions | 6 months
  Size and types of the lesions were examined at the beginning of treatment, and then after 2 weeks, 1, 3, and 6 months of therapy.
  Score 5 = white striae with erosive area more than I cm Score 4 = white striae with erosive area less than 1 cm Score 3 = white striae with atrophic area more than I cm Score 2 = white striae with atrophic area less than I cm Score I =mild white striae, no erythematous area Score 0 = no lesion, normal mucosa
Pain score (Visual analogue scale (VAS)), | 6 months
  Pain score was recorded at the beginning of treatment, and then after 2 weeks, 1, 3, and 6 months of therapy.
  Scale 0: no pain: VAS=0 Scale 1: mild pain: 0< VAS≤3.5 Scale 2: moderate pain: 3.5 <VAS≤7 Scale 3: severe pain: 7< VAS≤10.
Recurrence of disease | 3 months
  Recurrence within the following 3 months was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Enas Elgendy, ph.D, Principal Investigator — October 6 University
Locations (1):
- October 6 University, Cairo, Egypt